CLINICAL TRIAL: NCT04166266
Title: National Cohort of Patients Co-infected With Hepatitis B and Delta Viruses
Acronym: HEPDELTA
Status: Recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS HD EP01-HEPDELTA
Record Dates: First submitted 2019-09-12; First posted 2019-11-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis D, Chronic; Hepatitis B, Chronic
Keywords: safety; efficacy; evolution; treatment
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis B, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with co-infection with hepatitis B and Delta viruses,: Blood sampling for the biobank and, in addition, as sub-studies are planned on sub-groups of patients, additional blood samples are planned for the patients in these sub-studies.
  Interventions: Other: Blood draw for the laboratory assessment

INTERVENTIONS:
Other: Blood draw for the laboratory assessment — Blood sampling for the biobank and, in addition, as sub-studies are planned on sub-groups of patients, additional blood samples are planned for the patients in these sub-studies.

SUMMARY:
This is a multicentre observational study with prospective and retrospective data collection and retrospective data collection and biological collection from patients with HBV/HDV co-infection.

DETAILED DESCRIPTION:
This is an observatory for patients co-infected with hepatitis B and Delta viruses. Patients will be monitored according to the usual recommendations, depending on their status:

* Patients who have never received specific treatment for hepatitis Delta (untreated or receiving treatment with peginterferon alpha 2a alone) will be monitored according to current recommendations, once every 6 months;
* Patients treated or having been treated with a specific hepatitis Delta treatment will be monitored according to the compassionate access protocol or according to the recommendations of the AMM during treatment and according to routine follow-up after the end of treatment.

Participation in research entails the following additional procedures for patients, for each line of treatment, where applicable:

* Samples for the biobank,
* Self-administered questionnaires.

In addition, as sub-studies are planned on sub-groups of patients, these sub-studies may involve additional constraints/interventions

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Presenting a chronic HDV infection (positive serology),
* Who gave his written informed consent before any intervention and the day of inclusion at the latest,
* Affiliated to Health Insurance or to the "Aide Médicale d'Etat" (request for exemption pending).

Exclusion Criteria:

* Patient participating in another biomedical research with an exclusion period ongoing at inclusion,
* Vulnerable patient (minor, adults legally protected: under judicial protection, guardianship, or supervision, persons deprived of their liberty).
* Patients with predictable difficulties of follow-up according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients followed in the participating centers for their HBV/HDV co-infection are susceptible to be included.
  Patients who already started a specific treatment for their HDV infection will be included retrospectively, after they have signed an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
To study the natural or treated history of patients infected with HDV according to different management modalities. | At the end of the follow-up, december 2027
  This is a cohort in which many events will be studied. As the objectives are multiple, no primary endpoint has been defined.

SECONDARY OUTCOMES:
Number of patient's reported outcomes measured with specific questionnaire | weeks 24, 48, end of treatment and 48 weeks after the end of treatment
Quality of observance measured with specific questionnaire | weeks 24, 48, end of treatment and 48 weeks after the end of treatment
Alcohol consumption (AUDIT-c), tobacco and cannabis use | weeks 24, 48, end of treatment and 48 weeks after the end of treatment
Socio-economic situation measured with specific questionnaire | weeks 24, 48, end of treatment and 48 weeks after the end of treatment
Quality of life level measured with short-form 12 (SF12) questionnaire | At weeks 24, 48, end of treatment and 48 weeks after the end of treatment
Rate of patients achieving HBV DNA indetectability | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of early discontinuation of treatment due to an adverse event | At weeks 12, 24, 48, end of treatment
HDV RNA level | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
HDV RNA variation rate | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Breakthrough rate | At weeks 8, 12 and through the end of treatment (average 3 years)
Rate of sustained virological response | At weeks 12, 24, 36 and 48 and through the end of treatment (average 3 years)
  HDV RNA undetectability
Rate of partial virological response | At weeks 4, 8, 12 and through the end of treatment (average 3 years)
  reduction in Delta RNA of at least 2 log10 compared with the basal value, without undetectability
Rate of patients achieving HBs seroconversion | At weeks 12, 24, 48,through the end of treatment (average 3 years), and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Virological response delay | At weeks 8, 12 and through the end of treatment (average 3 years)
Number of different HDV resistance variants | Through treatment period, average 3 years
Number of patients with at least one resistance variant | Through treatment period, average 3 years
Fibrosis level | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of adverse event | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Death rate | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Liver transplantation rate | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Number and characterization of associated treatment with analogs and/or interferon | At weeks 4, 8, 12 and through the end of treatment (average 3 years
Rate of patients presenting an evolution towards hepatocellular carcinoma | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of patients presenting an evolution towards cirrhosis | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
  in non-cirrhotic patients
Rate of patients presenting a decompensated cirrhosis | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
  in non-cirrhotic patients
Change in HBs Ag from baseline | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of biochemical response | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
  Biochemical response is defined as ALT and aspartate aminotransferase (AST) normalization
Rate of patients achieving hepatitis B e (HBe) Ag negativation in patient initially HBeAg- positive | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of patients with appearance of anti-HBe Ab | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of patients achieving HBe seroconversion | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of spontaneous virological recovery | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
  Prolonged HDV RNA undetectability
Rate of patients achieving HBs Ag negativation | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)
Rate of patients with appearance of anti-HBs Ab | At weeks 12, 24, 48, end of treatment and 12, 24, 36 weeks after the end of treatment and every 24 weeks through study completion (max december 2027)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ZOULIM, Study Director — Hôpital de la Croix-Rousse
Locations (38):
- France (38):
  - CHU of Angers, Angers
  - Centre Hospitalier de la région annécienne, Annecy
  - Avicenne Hospital - Hepatology, Bobigny
  - Avicenne Hospital, Bobigny
  - Haut Lévêque Hospital, Bordeaux
  - Estaing Hospital, Clermont-Ferrand
  - Beaujon Hospital, Clichy
  - Centre Hospitalier Intercommunal, Créteil
  - Henri Mondor Hospital, Créteil
  - Bocage Hospital, Dijon
  - Michallon Hospital, Grenoble
  - Claude Huriez Hospital, Lille
  - Dupuytren Hospital, Limoges
  - Croix Rousse Hospital, Lyon
  - Edouard Herriot Hospital, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - SAint Joseph Hospital, Marseille
  - Saint Eloi Hospital, Montpellier
  - Hotel Dieu Hospital, Nantes
  - Hôtel-Dieu Hospital, Nantes
  - l'Archet 2 Hospital, Nice
  - La Source Hospital, Orléans
  - Bichat-Claude Bernard Hospital, Paris
  - Cochin Hospital, Paris
  - Hôpital Tenon, Paris
  - La Pitié Salpêtrière Hospital, Paris
  - Lariboisière Hospital, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Saint Antoine Hospital, Paris
  - Saint Louis Hospital, Paris
  - Saint-Antoine Hospital, Paris
  - Pontchaillou Hospital, Rennes
  - Charles Nicolle Hospital, Rouen
  - Nouvel Hôpital Civil, Strasbourg
  - Hôpital Rangueil, Toulouse
  - Rangueil Hospital, Toulouse
  - Trousseau Hospital, Tours
  - Paul Brousse Hospital, Villejuif

IPD SHARING:
Plan to Share IPD: No